CLINICAL TRIAL: NCT06557759
Title: The Effect of Listening to 30-Minutes of Calming Music on Mental Health Professionals
Brief Title: 30-Minutes of Listening to Calming Music on Attendees of a Workshop Session at a Local Conference
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Conference canceled due to hurricane
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB202401167
Record Dates: First submitted 2024-08-06; First posted 2024-08-16 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Depression; Anxiety; Autonomic Dysregulation
Keywords: Polyvagal Theory; Trauma; Adversity; Anxiety; Depression; Mental Health; Emotional Health; Music; Social Connection; Embodiment; Autonomic Reactivity; Body Sensations; Relaxation
MeSH Terms: conditions — Depression; Anxiety Disorders; Primary Dysautonomias; Wounds and Injuries; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The participants will listen to the brief music demo together after completing the pre-assessment. After the demo is completed, participants will listen to the 30-minutes of music. For those who opt out of listening to the 30-minutes of music, they will be asked to complete the post-assessment as they exit. Following the 30-minute music session, the remaining participants will be asked to complete the post-assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music (Experimental): Participants will be asked to listen to the brief music demo and the 30-minute music session. The pre- and post-assessments will require participants to complete a 5-10-minute online survey.
  Interventions: Behavioral: Listening to Calming Music

INTERVENTIONS:
Behavioral: Listening to Calming Music — Participants will listen to calming music, which may enhance health and wellness by reducing autonomic reactivity and improving bodily awareness, brain-body connection, and emotional wellbeing.

SUMMARY:
The goal of this clinical trial is to explore possible benefits and mechanisms through which listening to music can improve health and wellness. The main goals of the study are:

* To investigate whether pre-survey measures of autonomic reactivity relate to the overall functioning of participants.
* To examine the immediate effects of listening to the music.
* To identify individual characteristics that influence the immediate effects of listening to the music.

Participants will:

* complete the online pre-assessment measures assessing their adversity history, psychiatric symptomatology, autonomic reactivity, embodiment, and perceived social connection.
* Listen to the brief music demo
* Listen to the full 30-minute music session.
* Complete the online post-assessment measures assessing psychiatric symptomatology, autonomic reactivity, embodiment, and perceived social connection.

DETAILED DESCRIPTION:
It is the specific intent of this proposal to experimentally explore the possible benefits and mechanisms through which listening to the music can influence emotional health, embodiment, and autonomic functioning. This will be accomplished by our team by using well-validated self-report measures of mental health and autonomic reactivity.

Specific Aims:

Specific Aim 1: To investigate whether pre-intervention measures of ANS reactivity relate to the overall functioning of the participants.

•We will examine measures of autonomic reactivity to prior mental health and medical adversity, embodiment, and emotional and physical health.

Specific Aim 2: To identify the immediate effects of listening to the music •We will explore whether listening to the music leads to improvements in the functioning. First, we will compare the participants who opted to leave after the brief music demonstration to the participants who stayed for the additional 30-minutes of music. Next, we will focus on improvements following listening to the music.

Specific Aim 3: To identify individual characteristics that influence the effectiveness of listening to the music immediately

•We will explore the impact of specific vulnerability and resiliency factors (e.g., prior mental and medical adversity) on how well mental health providers benefit from listening to the music immediately.

Experimental design

* Participation is limited to those attending the Global Exchange Conference
* The participants will complete pre- and post-assessments that involve online measures.
* Music will be provided first in a brief music demo and then again in a 30-minute session.
* Between-subject analyses will compare those who listened only to the brief demo and withdrew participation against those who remained and listened to the 30-minutes of music to determine if those who listened to the 30-minutes of music exhibit greater improvements than those who did not. Within-subject analyses will determine the potential benefits of listening to the music for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 89
* Proficient in English
* Attendees of an online workshop session at the Global Exchange Conference

Exclusion Criteria:

* Over the age of 89

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-08 (Estimated); Primary Completion 2024-11-09 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Measuring Change in Autonomic Reactivity using the Body Perceptions Inventory Short Form | From baseline through study completion, an average of 1 day
  This 20-item measure is scored on a 5-point Likert scale (never = 1, occasionally = 2, sometimes = 3, usually = 4, always = 5). Items are summed to determine total autonomic reactivity score, with the higher scores indicating greater autonomic reactivity
Measuring change in Body Sensations using the Neuroception of Psychological Safety Scale | From baseline through study completion, an average of 1 day
  This 8-item body sensations subscale is scored on a 5-point likert scale. Items are summed together to create a total subscale, with higher scores relecting internal sensations of the body in a state of calm capturing the feelings of relaxation in the face and the body, steady heartbeat and breath, and settled stomach.
Assessing the Impact of Adversity History on the Effectiveness of Listening to Music | Baseline
  This measure assesses the impact of six types of traumatic experiences (childhood adverse experiences, childhood maltreatment, intimate partner maltreatment, other person maltreatment, life-threatening situations, sudden losses, and person health situations). Each item is scored on a 5-point Likert scale (did not occur = 0, occurred and no impact on my life = 1 to big impact on my life = 4). Items are summed to determine total impact scores.

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes P Dale, PhD, Principal Investigator — UF College of Medicine Jacksonville, Department of Psychiatry

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to protect the privacy of participants.

REFERENCES:
- [Background] Dale LP, Davidson C, Kolacz J. (2020). The Adverse and Traumatic Experiences Scale.
- [Background] Cabrera A, Kolacz J, Pailhez G, Bulbena-Cabre A, Bulbena A, Porges SW. Assessing body awareness and autonomic reactivity: Factor structure and psychometric properties of the Body Perception Questionnaire-Short Form (BPQ-SF). Int J Methods Psychiatr Res. 2018 Jun;27(2):e1596. doi: 10.1002/mpr.1596. Epub 2017 Nov 28. PMID 29193423
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Morton L, Cogan N, Kolacz J, Calderwood C, Nikolic M, Bacon T, Pathe E, Williams D, Porges SW. A new measure of feeling safe: Developing psychometric properties of the Neuroception of Psychological Safety Scale (NPSS). Psychol Trauma. 2024 May;16(4):701-708. doi: 10.1037/tra0001313. Epub 2022 Jul 18. PMID 35849369
- [Background] Kroenke, K., & Spitzer, R. L. (2002). Patient Health Questionnaire-8 (PHQ-8)